CLINICAL TRIAL: NCT04817137
Title: Validation of a Novel Non-invasive Continuous Blood Pressure Monitor in Children Ages 2- 17 Years-old
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: CareTaker Medical LLC (Industry)
Responsible Party: Principal Investigator, Karen Boretsky, Anesthesiologist, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-P00037138
Record Dates: First submitted 2021-03-16; First posted 2021-03-26 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All Enrolled Patients (Other): Patients will wear the Caretaker Pulse Decomposition Analysis (PDA) Device, which will record the patient's blood pressure.
  Interventions: Device: CareTaker PDA Device

INTERVENTIONS:
Device: CareTaker PDA Device — Non-invasive blood pressure monitoring

SUMMARY:
This is a prospective observational study to investigate if a non-invasive blood pressure monitoring device, the CareTaker Pulse Decomposition Analysis (PDA), can accurately measure blood pressure in children when compared to an arterial line. Enrolled patients will have the CareTaker PDA device placed on their finger during their operation to collect data for 30 minutes. Blood pressure readings from the CareTaker PDA device will be compared to measurements from the patient's indwelling arterial line, which will be placed as part of the patient's clinical care plan.

ELIGIBILITY:
Inclusion Criteria:

* Plan to receive an invasive arterial blood pressure monitor as part of their anesthesia care plan at the BCH Longwood campus

Exclusion Criteria:

* Patients with vascular or congenital heart disease known to affect large and small arteries
* Patients who declined to participate.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Comparison | One hour during procedure
  The accuracy of blood pressure measurements taken from the non-invasive blood pressure device will be compared to measurements taken from the patient's indwelling arterial line, which will be place as part of standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Boretsky, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hopsital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scheer B, Perel A, Pfeiffer UJ. Clinical review: complications and risk factors of peripheral arterial catheters used for haemodynamic monitoring in anaesthesia and intensive care medicine. Crit Care. 2002 Jun;6(3):199-204. doi: 10.1186/cc1489. Epub 2002 Apr 18. PMID 12133178
- [Background] Gratz I, Deal E, Spitz F, Baruch M, Allen IE, Seaman JE, Pukenas E, Jean S. Continuous Non-invasive finger cuff CareTaker(R) comparable to invasive intra-arterial pressure in patients undergoing major intra-abdominal surgery. BMC Anesthesiol. 2017 Mar 21;17(1):48. doi: 10.1186/s12871-017-0337-z. PMID 28327093
- [Background] Baruch MC, Kalantari K, Gerdt DW, Adkins CM. Validation of the pulse decomposition analysis algorithm using central arterial blood pressure. Biomed Eng Online. 2014 Jul 8;13:96. doi: 10.1186/1475-925X-13-96. PMID 25005686
- [Background] Phillips AA, Burr J, Cote AT, Foulds HJ, Charlesworth S, Bredin SS, Warburton DE. Comparing the Finapres and Caretaker systems for measuring pulse transit time before and after exercise. Int J Sports Med. 2012 Feb;33(2):130-6. doi: 10.1055/s-0031-1291185. Epub 2011 Nov 17. PMID 22095319
- [Background] The Handbook of Cuffless Blood Pressure Monitoring. Edited by J Sola, Delgado-Gonzalo R, 2019 Springer Nature Swirtzerland AG 2019.
- [Background] Heeney ND, Habib F, Brar GK, Krahn G, Campbell DA, Sanatani S, Claydon VE. Validation of finger blood pressure monitoring in children. Blood Press Monit. 2019 Jun;24(3):137-145. doi: 10.1097/MBP.0000000000000374. PMID 30840608
- [Background] Epstein S, Willemet M, Chowienczyk PJ, Alastruey J. Reducing the number of parameters in 1D arterial blood flow modeling: less is more for patient-specific simulations. Am J Physiol Heart Circ Physiol. 2015 Jul 1;309(1):H222-34. doi: 10.1152/ajpheart.00857.2014. Epub 2015 Apr 17. PMID 25888513
- [Derived] Boretsky KR, Nasr VG, Atkinson D, Baruch M. Comparison of continuous non-invasive blood pressure measurement using Vitalstream to invasive Intraarterial pressure in pediatric surgery. J Clin Anesth. 2025 Mar;102:111763. doi: 10.1016/j.jclinane.2025.111763. Epub 2025 Jan 23. PMID 39854999